CLINICAL TRIAL: NCT03460223
Title: Phase 1 Clinical Trial Using Mesenchymal Stem Cell as Individualized Medicine to Evaluate the Safety and Efficacy in Kidney Fibrosis
Brief Title: Safety and Efficacy Study of Mesenchymal Stem Cell in Treating Kidney Fibrosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ling Lu, Principal Investigator, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJLT006
Record Dates: First submitted 2018-02-23; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Renal Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conventional plus MSC treatment (Experimental)
  Interventions: Biological: MSC

INTERVENTIONS:
Biological: MSC — conventional plus MSC or placebo treatment

SUMMARY:
In progressive kidney diseases, fibrosis represents the common pathway to end-stage kidney failure. The potential for stem cells to treat kidney failure was recently confirmed. Particularly, mesenchymal stem cell (MSC) has been demonstrated to protect kidney function and alleviating renal injury in these patients. Therefore, the investigators propose a hypothesis that MSCs (MSC) can also improve the disease conditions of kidney fibrosis patients, particularly reducing the decompensated conditions in these patients.

DETAILED DESCRIPTION:
Kidney fibrosis represents the common pathway to end-stage kidney failure.The potential for stem cells to treat kidney failure was recently confirmed. In particular, mesenchymal stem cell (MSC) transplantation has been applicated in the clinic for treat several human diseases such as GVHD, kidyney injury and displayed good tolerance and efficiency. The purpose of this study is to learn whether and how MSCs (MSC) can improve the disease conditions in patients with kidney fibrosis. This study will also look at safety in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Glomerular sclerosis ratio ≤ 50%.
3. Renal tubulointerstitial fibrosis ratio ≤ 50%.
4. Negative pregnancy test.
5. Moderately active disease under standard treatment.

Exclusion Criteria:

1. Severe infection and cardiovascular disease, shock, secondary liver disease and malignant tumor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
BUN | 24 months
  The evaluation of serum levels of BUN
Cr | 24 months
  The evaluation of serum levels of Cr
eGFR | 24 months
  The evaluation of serum levels of eGFR
Cystatin C | 24 months
  The evaluation of serum levels of Cystatin C
Urine protein | 24 months
  The evaluation of serum levels of Urine protein

SECONDARY OUTCOMES:
Hb | 24 months
  The evaluation of serum levels of Hb
Hct | 24 months
  The evaluation of serum levels of Hct
Ca | 24 months
  The evaluation of serum levels of Ca
P | 24 months
  The evaluation of serum levels of P
ALT | 24 months
  The evaluation of serum levels of ALT
PTH | 24 months
  The evaluation of serum levels of PTH
VitD | 24 months
  The evaluation of serum levels of VitD
ALB | 24 months
  The evaluation of serum levels of ALB
TC | 24 months
  The evaluation of serum levels of TC
TG | 24 months
  The evaluation of serum levels of TG

OTHER OUTCOMES:
Evaluation of renal fibrosis | 24 months
  The pathology decrease in grade of renal fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Tang, M.D, PH.D, Study Chair — Nanjing Medical University